CLINICAL TRIAL: NCT06569394
Title: A Randomized, Placebo Controlled Study of Cannabidiol in Young Adult Cannabis Users
Brief Title: A Study of Cannabidiol in Young Adult Cannabis Users
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 23-0954; 1P50DA056408 (NIH)
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Cannabis Use Disorder

STUDY DESIGN:
Intervention Model Description: Double-blind placebo controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be blind to medication assignment, as will all care providers and investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Broad Spectrum Cannabidiol (bsCBD) 400 mg (Active Comparator): bsCBD in a 400 mg dose will be used as described in the study arms.
  Interventions: Drug: Broad Spectrum Cannabidiol (bsCBD) 400 mg
- Placebo (Placebo Comparator): A medically inert placebo medication will be used as described in the study arms.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Broad Spectrum Cannabidiol (bsCBD) 400 mg — Participants in this Arm will take 400 mg of bsCBD daily. Participants will take medication by mouth with food in the morning and evening.
  Arms: Broad Spectrum Cannabidiol (bsCBD) 400 mg
Drug: Placebo — Participants in this Arm will take a medically inert placebo. Participants will take medication by mouth with food in the morning and evening.
  Arms: Placebo

SUMMARY:
The investigators will study the harm-reducing effect of hemp-derived CBD in non-treatment-seeking emerging adults who use cannabis regularly. The study will use a novel naturalistic cannabis administration approach, which examines ecologically valid cannabis use utilizing a mobile lab setting to assess the effects of the cannabis products the participants regularly use. The investigators will recruit a sample of emerging adults, half of whom primarily use flower products and half of whom primarily use concentrate products. Individuals will be randomly assigned to hemp-derived CBD or placebo.

DETAILED DESCRIPTION:
Emerging adults have the highest prevalence of cannabis use and CUD of any age group. Despite high rates of use and CUD, treatment seeking is relatively uncommon among emerging adults. Those who use cannabis are less confident in their ability to abstain and show higher rates of ambivalence regarding the goal of abstinence than those who use other drugs. Thus, emerging adult cannabis users may be more receptive to non-abstinence or harm reduction approaches. The overarching aim of this proposal is to assess the effects of hemp-derived CBD in emerging adults on harms associated with cannabis use including subjective intoxication, affect and mood, psychotic experiences, and cognitive functioning, as well as to examine whether CBD supplementation reduces self-administration of THC and symptoms of CUD. The investigators propose a study design with high external validity and experimental controls to study the harm-reducing effect of hemp-derived CBD in non-treatment-seeking emerging adults who use cannabis regularly. The study will use a novel naturalistic cannabis administration approach, which examines ecologically valid cannabis use utilizing a mobile lab setting to assess the effects of the cannabis products the participants regularly use. The investigators will recruit a sample of emerging adults, half of whom primarily use flower products and half of whom primarily use concentrate products. Individuals will be randomly assigned to hemp-derived CBD or placebo, consistent with the preliminary studies that have approved US Food and Drug Administration (FDA) Investigation New Drug (IND 153535 and 157515).

The specific aims are to:

Aim 1: Test whether assignment to hemp-derived CBD, relative to placebo, over 8 weeks is associated with a) reduced self-administration of THC, b) a reduction in CUD symptoms, c) lower levels of anxiety, depression, d) better cognitive function, and e) higher anandamide (AEA) levels. Hypothesis: Compared to baseline, the CBD group will demonstrate reduced THC administration, fewer CUD symptoms, lower levels of anxiety and depression, and better cognitive functioning at 4 and 8 weeks compared to the placebo group. At 12 weeks (4 weeks post-trial), these effects will persist. Assignment to CBD will be correlated with higher AEA levels.

Aim 2: Test whether assignment to hemp-derived CBD, relative to placebo, reduces acute effects of cannabis administration on: a) subjective drug effects, b) cognitive function, and c) mood and psychotic symptoms. Hypothesis: Compared to cannabis self-administration at baseline (without CBD), the CBD group will demonstrate lower subjective drug effects (mood elevation, anxiety), fewer psychotic symptoms, and better cognitive functioning after cannabis self-administration at 4 and 8 weeks compared to the placebo group. At 12 weeks (4 weeks post-trial), these effects will persist.

Aim 3: Test whether cannabis product type (flower vs. concentrates) moderates the association between CBD assignment and a) cannabis use, b) mood and anxiety, and c) cognitive functioning in both longer-term (aim 1) and acute (aim 2) effects. Hypothesis: CBD effects will be greater among those who use concentrates compared to those who use flower products for both longer-term and acute effects.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-25
2. Must have used cannabis flower or concentrates at least five days per week for the past year.
3. Currently not seeking to cut down or stop cannabis use
4. At least two symptoms of a DSM-5 cannabis use disorder

Exclusion Criteria:

1. Use of any illicit substance besides alcohol, nicotine, or cannabis (e.g., cocaine, opiates, methamphetamine, MDMA, benzodiazepines, or barbiturates) in the past 60 days, as indicated by self-report and urine toxicology screening at the beginning of each study visit.
2. Alcohol use on 3 or more days per week, and/or >3 drinks per drinking day in the past 60 days. Participants must also have a breath alcohol level of 0 at the beginning of each study visit.
3. Daily nicotine use.
4. Meets DSM-5 diagnostic criteria for a psychotic disorder (e.g., schizophrenia, schizophreniform disorder, schizoaffective disorder), bipolar disorder, major depression with suicidal ideation, or a history of treatment for these disorders.
5. Current cardiovascular or respiratory disease (e.g., coronary artery disease, severe asthma, chronic obstructive pulmonary disease)
6. Current use of any psychotropic (e.g., antidepressants, anxiogenics) or hepatotoxic medication.
7. Current use of anti-epileptic medications (e.g., clobazam, sodium valproate) or medications known to have major interactions with Epidiolex (buprenorphine, leflunomide, levomethadyl acetate, lomitapide, mipomersen, pexidartinib, propoxyphene, sodium oxybate, and/or teriflunomide) or a history of seizures.
8. Current use of strong or moderate CYP3A4 inhibitors or inducers (commonly used examples not captured by other exclusion criteria include protease inhibitors, macrolide antibiotics [e.g., erythromycin], azole antifungals [e.g., ketoconazole], verapamil, and grapefruit juice).
9. Current use of strong or moderate CYP2C19 inhibitors or inducers (commonly used examples not captured by other exclusion criteria include proton pump inhibitors, prednisone, and norethisterone).
10. Current or past hepatocellular disease, as indicated by medical history or alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin greater than two times the upper limit of the normal range at screening.
11. For female participants, pregnancy or trying to become pregnant. A positive pregnancy test at the beginning of any study visit will result in exclusion from ongoing study participation.
12. For female participants, currently lactating.
13. For female patients of childbearing potential, not willing to use at least one approved method of birth control while taking the study medication, unless she is surgically sterile, partner is surgically sterile, or she is postmenopausal (one year).
14. Current suicidality risk as indicated during the conduct of the C-SSRS with concurrence after a study physician's or PI evaluation if the response to C-SSRS questions 1 or 2 is "yes"

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Difference in blood THC-COOH levels | 8 weeks
  THC-COOH levels in blood samples collected at baseline, Week 4, and Week 8 of medication ingestion.
Difference in blood THC levels | 1 hour pre and post THC self-administration at baseline, 4 weeks, and 8 weeks
  THC levels in blood samples collected before and after cannabis use at baseline, Week 4, and Week 8 of medication ingestion.
Difference in cannabis use | 8 Weeks
  Total number of days of cannabis use during the 8-week medication period as reported on daily diaries.

OTHER OUTCOMES:
Adverse effects | 8 weeks
  Adverse effects reported at Week 4 and Week 8 of medication ingestion
Difference in blood CBD levels | 8 weeks
  CBD levels in blood samples collected at Week 4 and Week 8 of medication ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Christian J Hopfer, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared through a NIDA P50 data sharing resource.